CLINICAL TRIAL: NCT04381104
Title: Effective Strategy to Cope the Pain and Discomfort Among Women Undergoing Mammography
Brief Title: Strategy to Cope Pain and Discomfort in Mammography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Anila Rahim, Anila Rahim, Dow University of Health Sciences
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: IRB-1391/DUHS/Approval/2019
Record Dates: First submitted 2020-05-07; First posted 2020-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Anxiety; Pain; Discomfort
Keywords: breast; mammography; paracetamol
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: This will be a 2 arms individual randomized controlled trial. The intervention arm will receive 2 capsules of paracetamols of 500mg while the control arm will receive 2 capsules of placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The hospital pharmacy department is involved in the development of identical medicines both paracetamol and placebo. Codings are done by the hospital pharmacy department and researchers including principal investigator, care provider, outcome assessor, and even participant will remain blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paracetamol (Active Comparator): Capsule Paracetamol 1000 mg 1 hour before the mammography procedure
  Interventions: Drug: Paracetamol
- Placebo (Placebo Comparator): The control arm will receive 2 capsules of placebo.
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Drug: Paracetamol — The intervention arm will receive 2 capsules of paracetamols of 500mg.
  Other Names: Panadol

SUMMARY:
Most of the women complain about the pain and discomfort during the mammography procedure. It is reported in the literature that most of the time these pain and discomfort are due to anxiety-related causes. During counseling before mammography scan, it was also observed that most of the women had a general belief that mammography is a very painful procedure and they have a negative perception about mammography. Thus, the Majority of pain seems due to anxiety-related issues. Studies also support this evidence and it is reported in the literature that most of the women avoid mammography scans due to this negative perception which causes delay and ultimately a late diagnosis.

To validate the exact nature of pain and discomfort during mammography and to find out the strategy to cope with this anxiety-related pain and discomfort, there is a dire need for a study that can address this problem. Additionally, in our setup, most of the women who came for mammography are illiterate and belonged to the low socio-economic status. In these women, due to the negative perception, refusal or withdrawal rate is higher for mammography scans.

A thorough literature search has revealed studies on this issue are scarce both nationally and internationally. In the current study, Paracetamol will be used as a possible intervention which is the safest premedication for reducing pain while achieving standard compression which is necessary for good image quality. Thus, this study can help develop a strategy to control mammography discontinuation due to pain and discomfort.

DETAILED DESCRIPTION:
Mammography is considered a fundamental part of diagnosis in modern health care services. It provides low dose soft tissue imaging of normal structure and pathology within the breast. A mammogram can be performed on both asymptomatic and symptomatic women with palpable lumps and any other complaints. It is an appropriate source of early detection for breast cancer in diagnostic imaging. This screening practice is associated with a strong reduction in mortality in breast cancer as many guidelines have already published. Thus, Mammography has been demonstrated as a "Gold Standard" technique used for Breast cancer Imaging.

Besides, a strong reliance on Mammographic examination that most of the females may experience breast pain and discomfort while achieving standard compression in mammography which is necessary for optimal image quality a number of trials have been published. Moreover, previously reported that anxiety-related psychological pain, false perception or fear of discomfort is a factual reason for pain and discomfort while performing mammography. Breast pain is also associated with the menstrual cycle and noncyclic (trauma, surgery, and infection). Although, pain, discomfort, anxiety and false beliefs is a major reason to discontinue this procedure and over the past decades taking part in mammography is quite challenging for many women.

Premeditated mammography with the aid of analgesics is one of the most suitable interventions for diminishing pain. In this current study, paracetamol is used as an intervention for diminishing pain during mammography. Previously, a study declared that paracetamol can reduce mild pain and most people can take this medicine safely. We planned this study to evaluate the effective strategy to cope with the pain and discomfort among women undergoing mammography.

ELIGIBILITY:
Inclusion Criteria:

* All females patients aged above 40 years attending Dow Radiology Department for Mammographic Examination for the first time as screening or diagnostic purposes

Exclusion Criteria:

* Patients in whom additional projections such as cone compression, magnification, axillary, cleavage projection, and extended views will be acquired.
* Post-operative cases
* Women already have painful tender breast lumps.
* Patient who are unable to cooperate with us to take medication (either placebo/paracetamol)
* Patient who haven't agreed to give informed consent
* Any prior history of Paracetamol reaction and toxicity
* Lactating mothers
* Females with the previous history of mammography exam

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 632 (Estimated)
Dates: Start 2019-11-21 (Actual); Primary Completion 2020-09-14 (Estimated); Study Completion 2020-11-20 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of paracetamol before performing mammography in reducing pain and discomfort during mammography procedure | 1 hour post medication
  The pain score is being assessed via visual analogue scale (VAS) in the two groups, i.e. paracetamol and placebo, before performing mammography

CONTACTS AND LOCATIONS:
Overall Officials: Anila Rahim, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dow Institute of Radiology, Dow University of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Freitas-Junior R, Martins E, Metran-Nascente C, Carvalho AA, Silva MFD, Soares LR, Ximenes CA. Double-blind placebo-controlled randomized clinical trial on the use of paracetamol for performing mammography. Medicine (Baltimore). 2018 Mar;97(13):e0261. doi: 10.1097/MD.0000000000010261. PMID 29595685
- [Derived] Rahim A, Rasheed B, Adil SO, Naz N, Aslam N. Effective strategy to cope the pain and discomfort among women undergoing mammography - A randomized controlled trial. Pak J Med Sci. 2023 Sep-Oct;39(5):1422-1428. doi: 10.12669/pjms.39.5.7500. PMID 37680791